CLINICAL TRIAL: NCT00661284
Title: A Study to Investigate the Duration of Maintained Efficacy in Patients With Rheumatoid Arthritis Who Had Treated With MRA
Brief Title: A Study of Duration of Maintained Efficacy in Rheumatoid Arthritis (RA) Patients Off Treatment With MRA(a Development Code of Tocilizumab, an Anti IL-6 Receptor Monoclonal Antibody.)
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: MRA226JP
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ⅰ: Subject who have participated in previous studies and achieved DAS28 of < 3.2 at the last observation and at least one time point among the two previous assessment time points in a previous studies.

SUMMARY:
A 52-week follow up study to investigate the duration of maintenance of efficacy in patients with RA and achieved low disease activity in clinical trials of MRA and stopped the treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients who achieved DAS28 of < 3.2 at the last observation and at least one time point among the two previous assessment time points in a previous studies.

Exclusion Criteria:

* Patients who receive DMARDs or immunosuppressants between the last observation in a previous studies and the first observation in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject who have participated in previous studies
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who maintained efficacy during 52-weeks after the last infusion of MRA in the previous studies. | every 4th week up to the 48th week
Relationship between serum IL-6 concentration at the last observation of the previous studies and the duration of maintenance of efficacy | throughout study

SECONDARY OUTCOMES:
Efficacy: Proportion of patients who maintained efficacy among patients whose DAS28 was <2.6 at the last observation of the previous studies. | throughout study
Efficacy: Time course of DAS28 during the treatment-free period in the present study | throughout study
Efficacy: Relationship between serum IL-6 concentration at the last observation of the previous studies and the time course of DAS28 during the treatment-free period in the present study. | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kimura, Study Chair — Chugai Pharmaceutical,Clinical Research Department 1
Locations (5):
- Japan (5):
  - Chugoku region, Chugoku
  - Kanto region, Kanto
  - Kyushu region, Kyushu
  - Sikoku region, Sikoku
  - Tohoku region, Tōhoku